CLINICAL TRIAL: NCT04608552
Title: Effect of Myofunctional Therapy on Outcomes in Mild to Moderate Sleep Apnea
Brief Title: Effect of Myofunctional Therapy on OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D2651-R
Record Dates: First submitted 2020-10-20; First posted 2020-10-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Apnea; Myofunctional Therapy; Chronic Disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Myofunctional Therapy (Active Comparator): Active Myofunctional Therapy is comprised of five 30-minute weekly sessions for 4 weeks.
  Interventions: Behavioral: OMT Exercises
- Inactive Myofunctional Therapy (Sham Comparator): Sham MT will be comprised of recommendations for five 30-minute nasal breathing exercises each week, use of nasal lavage with application of 10ml of saline in each nostril two times per day.
  Interventions: Behavioral: Nasal Breathing Exercises; Other: Use of Nasal Lavage

INTERVENTIONS:
Behavioral: OMT Exercises — Oral and oropharyngeal exercises
  Arms: Active Myofunctional Therapy
Behavioral: Nasal Breathing Exercises — Nasal breathing exercises each week
  Arms: Inactive Myofunctional Therapy
Other: Use of Nasal Lavage — Use of nasal lavage with application of 10ml of saline in each nostril two times per day
  Arms: Inactive Myofunctional Therapy

SUMMARY:
The primary medical therapies for patients with Obstructive Sleep Apnea syndrome (OSA) require the use of medical devices on a nightly basis to help control breathing during sleep, which can be difficult for patients with mild-to-moderate disease. Because many patients use these therapies on a limited basis, or stop using them altogether, they continue to be at increased risk of the consequences of untreated OSA. Untreated and undertreated OSA compounds the risk of OSA consequences over time, particularly with increasing age and weight. Orofacial Myofunctional Therapy (OMT) takes a rehabilitative approach to OSA and is comprised of isotonic and isometric exercises that target the oral (e.g., tongue) and oropharyngeal (e.g., soft palate, lateral pharyngeal wall) to help restore normal breathing and airway patency at night while asleep. Should the study have positive findings, OMT could become an important alternative therapy for patients with mild-to-moderate disease because patients could utilize a therapy that improves their nighttime breathing through daytime exercises and without the need for a burdensome medical device.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effect of Orofacial Myofunctional Therapy in Veterans with mild-to-moderate sleep apnea. The main question to be answered is whether OMT improves measures of OSA severity, patient functional status, and OSA symptoms when compared to sham OMT.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate OSA
* Entry criteria are as inclusive as possible and operationalized as follows: age>18 years old
* Confirmed diagnosis of OSA
* Having chronic symptoms per screening symptom checklist
* Fluency in English
* Must be getting care the VA San Diego Healthcare System

Exclusion Criteria:

* Cognitive impairment sufficient to cause inability to complete the protocol (per medical chart review)
* Low health literacy
* Residence in a geographical area outside of San Diego County
* Fatal comorbidity (life expectancy <6 months as indicated by treating physician)
* Significant documented substance/chemical abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Apnea Hypopnea Index (AHI; measure of sleep apnea disease severity) | 3 months and 6 months
  Compare the change in AHI between OMT and inactive OMT groups over the follow-up time points. Higher AHI scores indicate increase sleep apnea disease severity.

SECONDARY OUTCOMES:
Change in Functional Outcomes of Sleep Questionnaire (FOSQ; measure of daytime functioning) | 3 months and 6 months
  Compare the change in FOSQ between OMT and inactive OMT groups over the follow-up time points. Higher FOSQ scores indicate improved levels of daytime functioning.
Change in Epworth Sleepiness Score (ESS; measure of sleepiness) | 3 months and 6 months
  Change in ESS between OMT and inactive OMT groups over the follow-up time points. Higher ESS scores indicate higher sleepiness levels.
Change in Pittsburgh Sleep Quality Index (PSQI; measure of sleep quality) | 3 months and 6 months
  Change in PSQI between OMT and inactive OMT groups over the follow-up time points. Higher PSQI scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Stepnowsky, Jr., PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT04608552/ICF_000.pdf